CLINICAL TRIAL: NCT04336397
Title: Randomized Controlled Trial of the Stool DNA Test to Improve Colorectal Cancer Screening Among Alaska Native People
Brief Title: Stool DNA to Improve Colorectal Cancer Screening Among Alaska Native People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alaska Native Tribal Health Consortium (Other)
Collaborators: Mayo Clinic (Other); Yukon Kuskokwim Health Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1R01CA247642-01 (NIH)
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Results first posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Intervention Model Description: 3-arm cluster-randomized controlled trial
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- High Intensity (Active Comparator): Navigated tribal health worker telephone outreach up to 5 telephone calls and 1 mailed culturally appropriate educational material describing CRC screening options available. If MT-sDNA selected, sent a MT-sDNA kit and follow-up reminders.
  Interventions: Diagnostic Test: Multi-target stool DNA test; Diagnostic Test: Colonoscopy
- Medium Intensity (Active Comparator): 1 mailed culturally appropriate educational material describing CRC screening options available and 1 telephone call from a tribal health worker. If MT-sDNA selected, sent a MT-sDNA kit and follow-up reminders.
  Interventions: Diagnostic Test: Multi-target stool DNA test; Diagnostic Test: Colonoscopy
- Usual Care (No Intervention): usual care (i.e., opportunistic screening recommendation at a clinic visit)

INTERVENTIONS:
Diagnostic Test: Multi-target stool DNA test — Cluster randomized trial of high and medium intensity outreach with MT-sDNA or colonoscopy compared with usual care
  Other Names: Cologuard
  Arms: High Intensity; Medium Intensity
Diagnostic Test: Colonoscopy — Cluster randomized trial of high and medium intensity outreach with MT-sDNA or colonoscopy compared with usual care
  Arms: High Intensity; Medium Intensity

SUMMARY:
Only 59% of Alaska Native people have been adequately screened for colorectal cancer (CRC) despite having the highest reported incidence of CRC in the world. A new at-home multi-target stool DNA screening test (MT-sDNA; Cologuard®) with high sensitivity for pre-cancerous polyps and CRC is now available. MT-sDNA has not been tested for feasibility or acceptability within the Alaska tribal health care delivery system, and it is unknown whether use of this new test will increase Alaska Native CRC screening rates. The long-term study goal is to improve screening and reduce CRC-attributable mortality. The objective of this application is to test the effectiveness of MT-sDNA for increasing CRC screening in Alaska Native communities using a mixed methods, community-based participatory research (CBPR) approach. The study will be conducted in collaboration with regional Tribal health organizations responsible for providing health care to geographically remote Alaska Native communities. Although the proposed implementation strategy is evidence-informed and promising, it is novel in that MT-sDNA has not been evaluated in the tribal health setting or among rural/remote populations. Using the RE-AIM Model, the research will be multi-level, examining influence on patients, providers, and tribal health organizations (THOs). This research study will pursue two specific aims: (1) Identify patient-, provider-, and system-level factors associated with CRC screening preferences, uptake, and follow-up; and (2) test the effectiveness of graded intensity MT-sDNA intervention in the Alaska Native community setting. For the first aim, focus groups with Alaska Native people who are not adherent to CRC screening guidelines and interviews with healthcare providers will be used to identify factors for future intervention. For the second aim, a three-arm cluster randomized controlled trial (high intensity with patient navigation, medium intensity with mailed reminders, usual care) will provide evidence on the MT-sDNA usefulness (MT-sDNA sample quality and neoplastic yield) as well as the first data on MT-sDNA follow up adherence rates in the Alaska Native population, which will inform plans to scale-up the intervention model. This research has the potential to sustainably improve public health by increasing CRC screening rates among a rural/remote tribal population as well as provide a model for other integrated health systems that provide care to high-risk or underserved populations in the U.S. and worldwide.

DETAILED DESCRIPTION:
The study will employ a cluster-randomized design, in which 32 communities within one Tribal health region will be randomized to one of the two study intervention conditions, matched by community size, with 14 communities in the control arm. All Alaska Native adults aged 45-75 due for colorectal cancer (CRC) screening within each community will be offered the same intervention. At least 770 participants will be recruited in at least 13 communities per study arm.

1. High Intensity Intervention: Participants will receive navigated tribal health worker outreach, a mailed MT-sDNA kit, mailed culturally appropriate educational material describing CRC screening options available and follow-up reminders
2. Medium Intensity Intervention: Participants will receive mailed culturally appropriate educational material describing CRC screening options available, including MT-sDNA, and navigated follow-up outreach reminders
3. Usual Care (Control arm): All other communities in the participating Tribal health region will serve as the reference group receiving usual care (i.e., screening recommendation at a clinic visit) Participants receiving the high intensity intervention are expected to have a 20% increase in screening uptake while those receiving medium intensity intervention will have a 10% increase in screening uptake over those receiving usual care. The study will also measure MT-sDNA sample quality and neoplastic yield in these remote Alaska Native communities. The investigators anticipate that the proportion of MT-sDNA tests meeting quality control standards will be the same as in the general US population (96%) and that pre-cancerous polyp detection rates at diagnostic post-MT-sDNA colonoscopy will exceed routine clinical practice rates in the general US population (52%-67%).

During and following the graded intensity intervention, the investigators will survey samples of patients to evaluate their awareness and response to the CRC screening intervention. The investigators will assess their perceived severity, perceived susceptibility, perceived benefits, perceived barriers, and self-efficacy relevant to CRC screening as well as measure the time-to-respond and screening method used. The study will use focus groups and key informant interviews to learn about factors associated with screening response. For the focus groups, AN people ages 45-75 who are unscreened or non-adherent to screening guidelines (colonoscopy within 10 years, sigmoidoscopy within five years, or fecal occult blood testing within preceding 12 months) will be invited to provide their views on barriers to and facilitators of screening, including barriers described in the literature and identified in the investigators previous work. Non-adherence will be identified through tribal medical records. Each focus group will last up to two hours, and will include 6-8 participants. All focus groups will be stratified by gender, and focus groups will be balanced so that approximately equal numbers of men and women are included in the analysis.

The investigators will also conduct a brief survey and key informant interviews (6-8 clinician interviews at each location) among community health aides, providers, and tribal health system administrators using validated measures of intervention feasibility, acceptability, and appropriateness to characterize provider- and system-level barriers and promotors to MT-sDNA implementation.

ELIGIBILITY:
Inclusion Criteria:

* Alaska Native adults eligible to receive health care through the Alaska Tribal Health System
* Active health system users with at least one Alaska Tribal Health System visit in the previous three years
* Due for colorectal cancer screening (have not had colonoscopy in past 10 years or fecal occult blood test in past 1 year or flexible sigmoidoscopy in past 5 years)

Exclusion Criteria:

* First-degree relative diagnosed with CRC at age 60 or younger
* History of familial adenomatous polyposis
* Hereditary non-polyposis CRC
* Previous colonoscopic evidence of inflammatory bowel disease, Crohn's disease, colorectal adenomas, or CRC
* Known history of colectomy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2029 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Diana Redwood, PhD, Principal Investigator — Alaska Native Tribal Health Consortium
Locations (1):
- Yukon-Kuskokwim Health Corporation, Bethel, Alaska, United States

IPD SHARING:
Plan to Share IPD: Yes
Pending Tribal approval, the final combined dataset can be shared as a completely de-identified dataset as defined by the Health Information Portability and Accountability Act and excluding any variable causing risk of identification due to small numbers.
Supporting Information: Study Protocol
Time Frame: 2025
Access Criteria: Interested investigators would be required to enter into a data sharing agreement with the Alaska Native Tribal Health Consortium that includes the following: 1) a commitment to follow the Tribal approval process from concept proposal to dissemination; 2) a commitment to using the data only for research purposes and not to identify any individual participant; 3) a commitment to securing the data using appropriate computer technology; and 4) a commitment to destroying or returning the data after analyses are completed.

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Community
Period: Overall Study
Arm/Group | High Intensity | Medium Intensity | Usual Care
Started | 746; 16 Community | 696; 16 Community | 587; 14 Community
Completed | 746; 16 Community | 696; 16 Community | 587; 14 Community
Not Completed | 0; 0 Community | 0; 0 Community | 0; 0 Community

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Intensity | Medium Intensity | Usual Care | Total
Number analyzed (Participants) | 746 | 696 | 587 | 2029
Age, Customized [Count of Participants; unit: Participants]
  45-54 | 338 | 321 | 311 | 970
  55-64 | 267 | 242 | 178 | 687
  65-75 | 141 | 133 | 98 | 372
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 303 | 274 | 239 | 816
  Male | 443 | 422 | 348 | 1213
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Alaska Native | 746 | 696 | 587 | 2029
Region of Enrollment [Number; unit: participants]
  United States | 746 | 696 | 587 | 2029
CRC screening test requested [Count of Participants; unit: Participants] — Population: At baseline, no participants had chosen a colorectal cancer screening test.

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer Screening by Study Arm
Description: Incident CRC screening episode defined as having at least one of the following within 1 year of follow-up after randomization and intervention: colonoscopy; MT-sDNA with a negative result; or MT-sDNA with a positive result followed by a colonoscopy within 1 year.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | High Intensity | Medium Intensity | Usual Care
Number analyzed (Participants) | 746 | 696 | 587
Participants | 205 | 165 | 32
Statistical Analysis 1: Comparison: High Intensity vs Medium Intensity; Test type: Superiority; p = 0.04, Chi-squared; Odds Ratio (OR) = 1.2, 95% CI 2-sided [1.0 to 1.5]
Statistical Analysis 2: Comparison: High Intensity vs Medium Intensity vs Usual Care; Test type: Superiority; p < 0.01, Chi-squared

2. Secondary Outcome: Test Requested (MT-sDNA or Colonoscopy)
Description: Test requested (MT-sDNA or colonoscopy) by intervention participants
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | High Intensity | Medium Intensity
Number analyzed (Participants) | 539 | 410
Participants
  MT-sDNA | 384 | 277
  Colonoscopy | 155 | 133

3. Secondary Outcome: MT-sDNA Diagnostic Follow-up
Description: Rate of positive MT-sDNA test follow up to diagnostic colonoscopy
Time Frame: 1 year
Population: This measure only includes participants who had an abnormal MT-sDNA test in either the high- and medium-intensity intervention arms and whether they received a follow-up colonoscopy. Usual care arm was not offered MT-sDNA and so is not included in this secondary outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | High Intensity | Medium Intensity
Number analyzed (Participants) | 37 | 20
Participants | 29 | 20

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: The period used for adverse event reporting was from baseline study enrollment to study completion for each participant, an average of 1 year, 6 months. No adverse events occurred for any participants.
Arm/Group | High Intensity | Medium Intensity | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/746 | 0/696 | 0/587
Serious Adverse Events (participants affected / at risk) | 0/746 | 0/696 | 0/587
Other Adverse Events (participants affected / at risk) | 0/746 | 0/696 | 0/587

LIMITATIONS AND CAVEATS:
This study was limited to a single population group located in one geographical region.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-14): https://cdn.clinicaltrials.gov/large-docs/97/NCT04336397/Prot_SAP_000.pdf